CLINICAL TRIAL: NCT04514861
Title: Effectiveness of Measuring Local Tissue Oxygen in Response to Induced Hemodynamic Changes With the Profusa's Wireless Lumee Oxygen Platform in Patients With Peripheral Artery Disease (PAD)
Brief Title: Monitoring Local Tissue Oxygen Changes Using the Wireless Lumee Oxygen Platform in Correlation to TcPO2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Profusa, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TP0139; 4R44HL131366-02 (NIH); CFDA Number: 93.837 (Other: U.S. Department of Health and Human Services)
Record Dates: First submitted 2020-07-27; First posted 2020-08-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Arterial Disease; Tissue Oxygen Monitoring; TcPO2
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Single-arm, non-randomized, effectiveness and performance study with confirmatory device in subjects with PAD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tissue Oxygen Dynamics with Lumee Oxygen and TcPO2 (Other): Monitoring local subcutaneous tissue oxygen dynamics using the Wireless Lumee Oxygen Platform in correlation to TcPO2 measurements in the arm and foot
  Interventions: Device: Wireless Lumee Oxygen Platform

INTERVENTIONS:
Device: Wireless Lumee Oxygen Platform — The Lumee Oxygen Platform is designed to monitor oxygen dynamics with a hydrogel placed in subcutaneous tissue

SUMMARY:
The purpose of this study is to monitor changes in local tissue oxygen levels in participants with Peripheral Artery Disease (PAD) using the Wireless Lumee Oxygen Platform. A transcutaneous oxygen pressure (TcPO2) device is used to show correlations in oxygen dynamics. Oxygen dynamics are induced by a pressure cuff and position maneuvers. Study participants will participate in the study for 12 months with six (6) planned visits over the course of the study.

The investigational device, the Wireless Lumee Oxygen Platform, consists of the Lumee Oxygen, a sterile soft injectable oxygen-sensitive hydrogel, designed to sense and report oxygen levels in the subcutaneous tissue. After initial insertion of the hydrogel in the subcutaneous tissue using the Lumee Pen (a sterile disposable injector device), tissue oxygen levels can be monitored continuously using the Lumee Patch (a non-invasive, non-sterile, wireless electronic device to collect, analyze and report tissue oxygen levels sensed by Lumee Oxygen Hydrogel) attached to the skin through the Lumee Patch Adhesive (designed to adhere the Lumee Patch). The Lumee Patch sends collected tissue oxygen data to the Lumee App which displays the collected data and operates up to four Lumee Patches.

ELIGIBILITY:
Inclusion Criteria:

A suitable candidate must meet the following criteria:

* Male or female must be ≥ 18 years of age
* Diagnosed with PAD, stable at time of enrollment, and may include prior stable lower extremity revascularization
* Has been informed of the nature of the study, agrees to its provisions, and has signed the informed consent form prior to any study related procedure
* Should plan to be available for all safety follow-up examinations at the investigational site
* Is aware that the Lumee™ Oxygen hydrogels are intended to stay in the tissue indefinitely
* Is aware that photos of injection sites and wound site will be taken, and videos may be recorded

Exclusion Criteria:

A candidate will be excluded from the study if any of the following criteria are met:

* PAD of Rutherford Classification 5 or 6 at time of enrollment
* Subject has an active infection
* Subject has an open wound on limb included in study
* Known history of keloids, excessive fibrosis during wound healing
* Known allergies to Lumee™ Oxygen hydrogel components, local anesthetic agents, suture materials, or severe skin allergies to adhesives
* Any skin or musculoskeletal condition or deformity limiting injection of the Lumee™ Oxygen hydrogel or preventing subsequent attachments of the Lumee™ Patch system
* Any skin modification in the area of injection that would potentially influence device performance (for example tattoos or scars)
* Previous amputation proximal to the digital level on the limb included in the study
* Significant venous insufficiency resulting in swelling of the lower leg, ankle or foot or chronic venous stasis changes (CEAP clinical score ≥ 3)
* Any condition that at the discretion of the investigator, physician or designee will impact the safety of the subject or the scientific integrity of the trial
* Female subjects of childbearing capacity (not surgically sterile or menopausal for ≥ 1 year)
* Participation in another clinical study, that would potentially interfere with the participation in this study
* Subject requires dialysis
* Subject is immunocompromised
* Subject has incompressible arteries tested by occlusion test in the arm
* Inability to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of subcutaneous oxygen dynamics measured by the Wireless Lumee Oxygen Platform and a TcPO2 device in the arm | At 2 days (±1 day) after injection and at 3 months (±14 days) after injection
  Correlation of measurements between subcutaneous tissue oxygen concentration expressed by the Lumee Oxygen Index (LOI; unitless; measured by the Wireless Lumee Oxygen Platform) and transcutaneous partial pressure of oxygen (TcPO2; mmHg; measured by the Periflux System 5000 or Periflux System 6000) in the arm during changes of oxygen induced by pressure cuff.

SECONDARY OUTCOMES:
Correlation of subcutaneous oxygen dynamics measured by the Wireless Lumee Oxygen Platform and a TcPO2 device in the foot | 1-14 days after hydrogel insertion
  Correlation of measurements between subcutaneous tissue oxygen concentration expressed by the Lumee Oxygen Index (LOI; unitless; measured by the Wireless Lumee Oxygen Platform) and transcutaneous partial pressure of oxygen (TcPO2; mmHg; measured by the Periflux System 5000 or Periflux System 6000) in the foot during changes of oxygen induced by pressure cuff.

OTHER OUTCOMES:
Correlation of subcutaneous oxygen dynamics measured by the Wireless Lumee Oxygen Platform and a TcPO2 device in the arm and foot | Throughout 12 months.
  Correlation of measurements between subcutaneous tissue oxygen concentrations expressed by the unitless Lumee Oxygen Index (LOI; measured by the Wireless Lumee Oxygen Platform) and transcutaneous partial pressure of oxygen (TcPO2; measured by the Periflux System 5000 or Periflux System 6000) in arm and foot during changes of oxygen induced by pressure cuff and positional maneuvers at various timepoints.
Occurrence of Adverse Events | Throughout 12 months and during all unscheduled visits
Lumee™ Patch and Lumee™ Oxygen hydrogel placement site skin observations | Throughout 12 months and during all unscheduled visits
  Skin observations will follow a grading system for Erythema, Edema and Hematoma at the injection site and the skin area where the Lumee Patches were adhered. The scores rank from 0= No Edema/Erythema/Hematoma, 1= very slight, 2 = well-defined, 3=moderate to 4= severe. Incidences of these ranks will we analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Lozano, PhD, Study Director — Profusa, Inc.
Locations (3):
- United States (3):
  - San Francisco General Hospital, San Francisco, California
  - San Francisco Veterans Affairs Medical Center (SFVAMC), San Francisco, California
  - UCSF Medical Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montero-Baker MF, Au-Yeung KY, Wisniewski NA, Gamsey S, Morelli-Alvarez L, Mills JL Sr, Campos M, Helton KL. The First-in-Man "Si Se Puede" Study for the use of micro-oxygen sensors (MOXYs) to determine dynamic relative oxygen indices in the feet of patients with limb-threatening ischemia during endovascular therapy. J Vasc Surg. 2015 Jun;61(6):1501-9.e1. doi: 10.1016/j.jvs.2014.12.060. PMID 26004327
- [Background] Chien JS, Mohammed M, Eldik H, Ibrahim MM, Martinez J, Nichols SP, Wisniewski N, Klitzman B. Injectable Phosphorescence-based Oxygen Biosensors Identify Post Ischemic Reactive Hyperoxia. Sci Rep. 2017 Aug 15;7(1):8255. doi: 10.1038/s41598-017-08490-0. PMID 28811566
- [Background] Wisniewski NA, Nichols SP, Gamsey SJ, Pullins S, Au-Yeung KY, Klitzman B, Helton KL. Tissue-Integrating Oxygen Sensors: Continuous Tracking of Tissue Hypoxia. Adv Exp Med Biol. 2017;977:377-383. doi: 10.1007/978-3-319-55231-6_49. PMID 28685468
- [Background] Nichols SP, Balaconis MK, Gant RM, Au-Yeung KY, Wisniewski NA. Long-Term In Vivo Oxygen Sensors for Peripheral Artery Disease Monitoring. Adv Exp Med Biol. 2018;1072:351-356. doi: 10.1007/978-3-319-91287-5_56. PMID 30178370
- [Background] Kanick SC, Schneider PA, Klitzman B, Wisniewski NA, Rebrin K. Continuous monitoring of interstitial tissue oxygen using subcutaneous oxygen microsensors: In vivo characterization in healthy volunteers. Microvasc Res. 2019 Jul;124:6-18. doi: 10.1016/j.mvr.2019.02.002. Epub 2019 Feb 8. PMID 30742844